CLINICAL TRIAL: NCT01983878
Title: A Phase 2 Study of Ramucirumab in the Treatment of Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma Following Disease Progression on First Line Platinum- or Fluoropyrimidine-Containing Combination Therapy in Japanese Patients
Brief Title: A Study of Ramucirumab in Treating Japanese Participants With Metastatic Gastric or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15045; I4T-JE-JVCL (Other: Eli Lilly and Company)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ramucirumab (Experimental): Ramucirumab 8 milligrams per kilogram (mg/kg) administered intravenously (IV) once every 2 weeks. Treatment will continue until there is evidence of progressive disease (PD), the development of unacceptable toxicity, protocol noncompliance or withdrawal of consent.
  Interventions: Drug: Ramucirumab

INTERVENTIONS:
Drug: Ramucirumab — Administered IV
  Other Names: LY3009806; IMC-1121B

SUMMARY:
The purpose of this study is to evaluate progression-free survival in participants with gastric or gastroesophageal junction cancer who have had disease progression following first-line therapy who undergo treatment with ramucirumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed gastric carcinoma, including gastric adenocarcinoma or Gastroesophageal Junction (GEJ) adenocarcinoma
* Metastatic disease or locally recurrent, unresectable disease
* Measurable disease and/or evaluable disease
* Experienced disease progression during or within 4 months after the last dose of first-line therapy for metastatic disease, or during or within 6 months after the last dose of adjuvant therapy
* Life expectancy of at least 3 months
* Resolution to Grade less than or equal to 1 by the National Cancer Institute Common Terminology Criteria for Adverse , Version 4.03, of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy
* Eastern Cooperative Oncology Group performance status score of 0-1
* Has adequate organ function
* Must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods), if sexually active
* Female participants of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to enrollment

Exclusion Criteria:

* Documented and/or symptomatic brain or leptomeningeal metastases
* Bone metastases
* Experienced Grade 3/4 gastrointestinal (GI) bleeding within 3 months prior to enrollment
* Experienced any arterial thromboembolic event within 6 months prior to enrollment
* Ongoing or active significant infection, symptomatic congestive heart failure (CHF), unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thromboembolic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the investigator
* Ongoing or active psychiatric illness or social situation that would limit compliance with study requirements
* Blood pressure in abnormal range despite standard medical management
* Has a serious or nonhealing wound, ulcer, or bone fracture
* Received chemotherapy, radiotherapy, immunotherapy, or targeted therapy for gastric cancer
* Received any investigational therapy within 30 days prior to enrollment
* Undergone major surgery within 28 days prior to enrollment, or subcutaneous venous access device placement within 7 days prior to enrollment
* Received prior therapy with an agent that directly inhibits vascular endothelial growth factor (VEGF) or vascular endothelial growth factor receptor 2 (VEGFR-2) activity (including bevacizumab), or any anti-angiogenic agent
* Receiving chronic therapy with nonsteroidal anti-inflammatory drugs or receiving other antiplatelet agents. Aspirin use at doses up to 325 milligrams per day is permitted
* Has elective or planned major surgery to be performed during the course of the clinical study
* Has a known allergy to any of the treatment components
* Pregnant or breastfeeding
* Have positive test results for human immunodeficiency virus, hepatitis B, or hepatitis C antibodies
* Known alcohol or drug dependency
* Previous or concurrent malignancy except for basal or squamous cell skin cancer (nonmelanoma) and/or pre-invasive carcinoma of the cervix, mucosal gastrointestinal or uterine carcinoma, or other solid tumors treated curatively and without evidence of recurrence for at least 3 years prior to enrollment
* Currently enrolled in a clinical trial involving an investigational product or non-approved use of a drug or device (other than the study drug/device used in this study), or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri from 9 AM to 5 PM Eastern Time (UTC/GMT-5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- Japan (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ehime
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hyōgo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shizuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Yamaguchi K, Fujitani K, Nagashima F, Omuro Y, Machida N, Nishina T, Koue T, Tsujimoto M, Maeda K, Satoh T. Ramucirumab for the treatment of metastatic gastric or gastroesophageal junction adenocarcinoma following disease progression on first-line platinum- or fluoropyrimidine-containing combination therapy in Japanese patients: a phase 2, open-label study. Gastric Cancer. 2018 Nov;21(6):1041-1049. doi: 10.1007/s10120-018-0811-4. Epub 2018 Mar 5. PMID 29508095

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant study completion was defined as participant assessment at the 12-week visit or withdrawal from the study.
Groups:
- Ramucirumab 8 mg/kg: Ramucirumab 8 milligrams per kilogram (mg/kg) administered intravenously (IV) once every 2 weeks. Treatment continued until there is evidence of progressive disease (PD), the development of unacceptable toxicity, protocol non-compliance, or withdrawal of consent.
Period: Overall Study
Arm/Group | Ramucirumab 8 mg/kg
Started | 36
Received At Least One Dose of Study Drug | 36
Completed | 36
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all enrolled participants who received at least one dose of the study drug.
Groups:
- Ramucirumab 8 mg/kg: Ramucirumab 8 mg/kg administered IV once every 2 weeks. Treatment continued until there is evidence of PD, the development of unacceptable toxicity, protocol non-compliance, or withdrawal of consent.
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  Japan | 36
Eastern Cooperative Oncology Group performance status (ECOG PS) 0 vs. 1 [Number; unit: Participants] — 0 = Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    Performance Status = 0 | 24
    Performance Status = 1 | 12
Basis for Pathological Diagnosis [Number; unit: Participants]
  Histopathological | 36
  Cytological | 0
Pathological Diagnosis [Number; unit: Participants]
  Adenocarcinoma, Gastroesophageal Junction | 1
  Adenocarcinoma, Gastric | 35
Initial Tumor Location [Number; unit: Participants]
  Body of stomach | 19
  Gastric Cardia | 3
  Gastric, Antrum | 14
Human Epidermal Growth Factor Receptor 2 (HER2) Status [Number; unit: Participants]
  Positive | 6
  Negative | 26
  Not Done | 3
  Unknown | 1
Grade [Number; unit: Participants]
  Well-differentiated (Low grade) | 4
  Moderately differentiated (Intermediate grade) | 11
  Poorly differentiated (High grade) | 20
  Not Applicable | 1
Histology [Number; unit: Participants]
  Intestinal | 15
  Diffuse | 13
  Mixed | 5
  Not Applicable | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Progression-Free at 12 Weeks (Progression-Free Survival [PFS] Rate at 12 Weeks)
Description: The 12-week PFS rate is the probability of participants who survived during the first 12 weeks in the study without disease progression. It was estimated using the Kaplan-Meier method for the main analysis of the 12-week PFS rate.
Time Frame: 12 Weeks
Population: Full Analysis Set (FAS): all enrolled participants who received at least one dose of the study drug. 8 participants were censored.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Ramucirumab 8 mg/kg: Ramucirumab 8 mg/kg administered IV once every 2 weeks. Treatment continued until there was evidence of progressive disease (PD), the development of unacceptable toxicity, protocol non-compliance, or withdrawal of consent.
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
Percentage of Participants | 23.8 [12.4 to 37.2]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: The time from baseline to measured Progressive Disease (PD) as defined by RECIST v.1.1 [defined as > 20% increase from smallest sum of longest diameter recorded since treatment started (best response)], or death due to any cause, whichever is first.
Time Frame: Baseline to Measured PD or Death from Any Cause (Up to 30.3 weeks)
Population: FAS: all enrolled participants who received at least one dose of the study drug. 8 participants were censored.
Measure: Median (90% Confidence Interval); unit: Weeks
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
Weeks | 6.6 [6.1 to 7.1]

3. Secondary Outcome: Percentage of Participants Achieving Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: Participants achieved an objective response if they had a best overall response of CR or PR. According to RECIST v1.1, PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter; CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all nontarget lesions, and the normalization of tumor marker levels [if tumor markers were initially above the upper limit of normal (ULN)]. The percentage of participants who achieved an objective response = (number of participants with CR or PR)/(number of participants assessed)*100.
Time Frame: Baseline to Measured PD or Death from Any Cause (Up to 38.0 Weeks)
Population: FAS: all enrolled participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
Percentage of Participants | 0 [0.00 to 7.98]

4. Secondary Outcome: Percentage of Participants Achieving Stable Disease (SD) or a Confirmed CR or PR [Disease Control Rate (DCR)]
Description: Participants achieved disease control if they had a best overall response of CR, PR or SD. According to RECIST v1.1, CR was the disappearance of all non-nodal target lesions, with the short axes of any target lymph node reduced to <10 mm, the disappearance of all non-target lesions, and the normalization of tumor marker levels (if tumor markers were initially above the ULN); PR was defined as at least a 30% decrease in the sum of the diameters of target lesions (including the short axes of any target lymph node), taking as reference the baseline sum diameter. SD was neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD, taking as reference the smallest sum diameter since treatment started. The percentage of participants who achieved disease control = (number of participants with CR, PR, or SD)/(number of participants assessed)*100.
Time Frame: Baseline to Measured PD or Death from Any Cause (Up to 12 Months)
Population: FAS: all enrolled participants who received at least one dose of the study drug.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
Percentage of Participants | 30.6 [18.18 to 45.47]

5. Secondary Outcome: Overall Survival (OS)
Description: The OS time is defined as the time from baseline to the date of death from any cause. If a participant is not known to have died on or before the date of data cut-off, OS data will be censored on the last date (on or before the cut-off date) the participant was known to be alive.
Time Frame: Baseline to Death from Any Cause (Up to 13 Months)
Population: FAS: all enrolled participants who received at least one dose of the study drug. 18 participants were censored.
Measure: Median (90% Confidence Interval); unit: Months
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
Months | 8.6 [5.7 to 10.7]

6. Secondary Outcome: Number of Participants With Anti-Ramucirumab Antibodies
Description: A sample will be considered positive for circulating anti-ramucirumab antibodies if it exhibits a post-baseline antibody level that exceeds the upper 95% confidence interval of the mean determined from the normal anti-ramucirumab level seen in healthy untreated individuals. A participant will be considered to have an anti-ramucirumab response if there are 2 consecutive positive samples or if the final sample tested is positive.
Time Frame: Cycle 1: Pre-infusion, Cycle 2: Pre-infusion, Cycle 3: Pre-infusion, Follow Up
Population: All enrolled participants who received at least one dose of study drug and had evaluable immunogenicity data.
Measure: Number; unit: participants
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 36
participants | 1

7. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Ramucirumab
Time Frame: Cycle 1 Day 1: Pre-Dose, End of Infusion. 1, 4, 23, 47, 95, 167, 263, and 335 Hours Post-Dose
Population: PK population: enrolled participants who received at least one dose of the study drug and had evaluable ramucirumab PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (μg/mL)
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 6
micrograms/milliliter (μg/mL) | 161 (16.2)

8. Secondary Outcome: PK: Area Under the Curve Time Zero to Infinity (AUC[0-∞]) of Ramucirumab
Time Frame: Cycle 1 Day 1: Pre-Dose, End of Infusion: 1, 4, 23, 47, 95, 167, 263, and 335 Hours Post-Dose
Population: as for outcome 7
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours x micrograms/milliliters (h*μg/mL)
Arm/Group | Ramucirumab 8 mg/kg
Number analyzed (Participants) | 6
hours x micrograms/milliliters (h*μg/mL) | 25600 (34.2)

ADVERSE EVENTS:
Arm/Group | Ramucirumab 8 mg/kg
Serious Adverse Events (participants affected / at risk) | 7/36
Other Adverse Events (participants affected / at risk) | 35/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab 8 mg/kg (N=36)
Ileus (Gastrointestinal disorders) | 2 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab 8 mg/kg (N=36)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Ascites (Gastrointestinal disorders) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 9 (16)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (5)
Stomatitis (Gastrointestinal disorders) | 2 (2)
Face oedema (General disorders) | 3 (3)
Fatigue (General disorders) | 3 (5)
Malaise (General disorders) | 6 (6)
Oedema (General disorders) | 2 (2)
Oedema peripheral (General disorders) | 5 (5)
Pyrexia (General disorders) | 4 (4)
Jaundice cholestatic (Hepatobiliary disorders) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (3)
Upper respiratory tract infection (Infections and infestations) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (5)
Platelet count decreased (Investigations) | 4 (4)
White blood cell count decreased (Investigations) | 3 (3)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Headache (Nervous system disorders) | 3 (4)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 7 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days